CLINICAL TRIAL: NCT01751269
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Single and Multiple-Dose Study of the Safety, Tolerability, Pharmacokinetics of Intravenous RPX7009 in Healthy Adult Subjects.
Brief Title: Safety, Tolerability, Pharmacokinetics of Intravenous RPX7009 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rempex Pharmaceuticals (a wholly owned subsidiary of The Medicines Company) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rempex 402
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Volunteers; Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — RPX7009; beta-Lactamase Inhibitors; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ascending Single and Multiple dose of RPX7009 (Experimental): Ascending Single and Multiple dose of RPX7009
  Interventions: Drug: RPX7009
- Normal Saline (Placebo Comparator): Ascending Single and multiple dose of normal saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RPX7009 — Ten (10) cohorts of 8 subjects (6 active and 2 placebo) are planned for evaluation.
  Other Names: (beta-lactamase inhibitor)
  Arms: Ascending Single and Multiple dose of RPX7009
Drug: Placebo — Ten (10) cohorts of 8 subjects (6 active and 2 placebo) are planned for evaluation.
  Other Names: Normal saline
  Arms: Normal Saline

SUMMARY:
RPX7009 (beta-lactamase inhibitor) is being studies in combination with a carbapenem biapenem to treat bacterial infections, including those due to multi-drug resistant bacteria.

DETAILED DESCRIPTION:
The worldwide spread of resistance to antibiotics among Gram-negative bacteria, particularly members of the ESKAPE group of pathogens, has resulted in a crisis in the treatment of hospital acquired infections. In particular, the recent dissemination of a serine carbapenemase (e.g., KPC) in Enterobacteriaceae in US hospitals now poses a considerable threat to the carbapenems and other members of the beta-lactam class of antimicrobial agents.

Rempex is developing a fixed combination antibiotic of a carbapenem plus a new beta-lactamase inhibitor (RPX7009) which has activity against serine beta-lactamases, including KPC. This Phase 1 study will assess the safety, tolerability and pharmacokinetics of RPX7009, administered alone, in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and/or females (of Non Child-bearing potential), 18 to 55 years of age
* Body mass index (BMI) ≥ 18.5 and ≤ 29.9 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive).
* Medically healthy with clinically insignificant screening results
* Non-tobacco/nicotine-containing product users for a minimum of 6 months prior to Day 1.
* Sexually abstinent or use acceptable methods of birth control

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* History or presence of alcoholism or drug abuse within the 2 years prior to Day 1.
* Documented hypersensitivity reaction or anaphylaxis to any medication.
* Use of any over-the-counter (OTC) medication, including herbal products and vitamins, within the 7 days prior to Day 1. Up to 2 grams per day of acetaminophen is allowed for acute events at the discretion of the PI.
* Plasma donation within 7 days prior to Day 1.
* Subjects who have any abnormalities on laboratory values at screening or check-in (Day -1).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety from baseline through the end of the study. | Study Day 1 to Day 13.
  Number of patients with adverse events; assessed by patient reporting, collection of vital signs, ECGs and absolute values and changes over time of hematology, chemistry and urinalysis.

SECONDARY OUTCOMES:
Composite of PK parameters RPX7009 & placebo following single dose administration. | Study Day 1 to Day 12
  Plasma AUC0-t, AUC0-inf, Cmax, and Tmax.

CONTACTS AND LOCATIONS:
Overall Officials: Jefferey Loutit, MBChB, Study Director — Sponsor GmbH
Locations (1):
- CMAX, Adelaide, South Australia, Australia

REFERENCES:
- [Derived] Griffith DC, Loutit JS, Morgan EE, Durso S, Dudley MN. Phase 1 Study of the Safety, Tolerability, and Pharmacokinetics of the beta-Lactamase Inhibitor Vaborbactam (RPX7009) in Healthy Adult Subjects. Antimicrob Agents Chemother. 2016 Sep 23;60(10):6326-32. doi: 10.1128/AAC.00568-16. Print 2016 Oct. PMID 27527080